CLINICAL TRIAL: NCT05481697
Title: Unintentional Weight Loss and Cancer: A Prospective Trial of Patient-centered Weight Tracking Combined With GRAIL Galleri Testing to Improve Early Detection
Brief Title: Unintentional Weight Loss and Cancer: A Prospective Trial of Patient-centered Weight Tracking Combin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: University Hospitals Seidman Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE3Y22
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Unintended Weight Loss
Keywords: GRAIL Galleri; Unintended Weight Loss; UWL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UWL and GRAIL Galleri Testing (Experimental): Enrolled participants will have an initial blood sample taken and record their weights weekly on a FitBit Aria scale for three years to detect for UWL
  Those who unintentionally lost lost ≥5% from their baseline weight will be identified and have a GRAIL Galleri blood test, physical examination, imaging, and cancer screenings to test for malignancy
  Interventions: Diagnostic Test: GRAIL Galleri

INTERVENTIONS:
Diagnostic Test: GRAIL Galleri — A blood test that aims to detect cancers earlier by looking for abnormal DNA shed from cancer cells into the blood.

SUMMARY:
Unintentional weight loss (UWL) is commonly associated with a wide variety of diseases and there is still no valid diagnostic pathway for evaluating UWL. When detecting UWL coupled with GRAIL Galleri testing, (an investigational pan-cancer early detection test), it is thought that there is a greater positive predictive value in detecting malignancies. This study aims to test the potential synergistic effects of UWL detection and GRAIL usage to detect malignancy at an even earlier rate. UWL will be measured using weekly weight tracking.

DETAILED DESCRIPTION:
Enrolled participants will be provided with a Fitbit Aria Smart Scale and will be asked to weigh themselves each week at a similar time of day wearing a similar amount of clothing for a total of three years. These weight data will be automatically pushed to the Fitbit cell phone application and patients who lost ≥5% from their baseline will be identified, and the intentionality of this weight loss (intentional or unintentional) will be assessed. All patients with UWL will be asked to have a GRAIL Galleri test, a health history and physical examination, a blood draw, imaging, routine cancer screenings done if not already completed, and referral to a specialist if a new cancer is detected.

ELIGIBILITY:
Inclusion Criteria:

* Age range: from 40 to 80 years
* Access to a device (cellphone, computer, tablet) that is compatible with the Fitbit Aria Air smart scale utilized in this study
* Willing to comply with all study procedures and be available for the duration of the study
* Subjects must be mentally competent and must have the ability to understand and the willingness to sign a written informed consent document
* Subjects must speak English to maximize chance of understanding the trial rational and study procedures

Exclusion Criteria:

* Active cancer diagnosis - current diagnosis, currently undergoing cancer treatment, or concluded cancer treatments within 3 years
* Actively trying to lose weight with medications or bariatric surgery
* Pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Malignant UWL Detection | Up to 3 years post-enrollment
  High-risk participant cohorts who have lost greater than or equal to 5% of their body weight at initial enrollment over the 3-year weight measuring period will be given a GRAIL Galleri test. If positive, the participant will be given laboratory work, imaging, and a physical examination to diagnose the malignancy.

SECONDARY OUTCOMES:
Non-Malignant UWL Detection | Up to 3 years post-enrollment
  Participants who have lost greater than or equal to 5% of their body weight at initial enrollment over the 3-year weight measuring period but tested negatively during a GRAIL Galleri test will be seen by a specialist to determine their underlying cause of UWL.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan M Winter, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States